CLINICAL TRIAL: NCT04710160
Title: Clinical and Radiographic Evaluation in Pulpotomy of Primary Molars Using Novel Fast-setting Calcium Silicate Cement (Protooth) Versus Mineral Trioxide Aggregate (MTA): A Pilot Study
Brief Title: Clinical and Radiographic Evaluation in Pulpotomy of Primary Molars Using Protooth Vs. MTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nashwa Ossama Ahmed Elshaer, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pedo193
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Clinical Evaluation Including Pain and Swelling
Keywords: Pulpotomy , Primary molars , Protooth , MTA
MeSH Terms: interventions — mineral trioxide aggregate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel fast setting calcium silicate ( Protooth) (Active Comparator): In the form of powder and liquid to be mixed together to form paste.
  Interventions: Drug: Novel fast-setting calcium silicate cement (Protooth)
- MTA (Experimental): In form of powder to be mixed with saline to form paste.
  Interventions: Drug: Novel fast-setting calcium silicate cement (Protooth)

INTERVENTIONS:
Drug: Novel fast-setting calcium silicate cement (Protooth) — In form of power and liquid to be mixed together to form a paste.
  Other Names: mineral trioxide aggregate (MTA )

SUMMARY:
The aim of the study is to evaluate the clinical and radiographic success in pulpotomy using novel fast-setting calcium silicate cement (Protooth) versus MTA in exposed primary molars.

ELIGIBILITY:
Inclusion Criteria:

* Complete physical and mental health, with no confounding history of systemic disease and/or use of special local or systemic drugs
* No allergic reactions recorded in patient history
* Having primary molar teeth in one jaw, having deep caries and vital pulp.
* No history of spontaneous pain, pathologic mobility, draining sinus tract, redness or swelling of vestibule
* Normal gingival and periodontal condition, with no sensitivity to vestibular palpation, and no pain on percussion test

  * Radiographic criteria:
* No sign of radiolucency in periapical or furcation area
* No widening of PDL space or loss of lamina dura continuity
* No evidence of internal/external pathologic root resorption

Exclusion Criteria:

* Lack of informed consent by the child patient's parent
* Lack of informed consent by the child patient's parent
* Unable to attend follow-up visits.
* Refusal of participation.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-10-22 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation including postoperative pain , pain on percussion or palpation will be measured using VAS | 12 months
  Post-operative pain following pulpotomy treatment will be measured.
  A pain chart using visual analogue scale (VAS) will be used to record the patients' pain levels. The VAS (0-10 scale) consists of a line anchored by two extremes "No pain" and "the worst pain". Patients will be asked to choose the mark that represented their level of pain from 0 to 10. Pain level will be assigned as follow:
  0, "no pain" 1-3, "mild pain" 4-6, "moderate pain" 7-10, "severe pain" Using the VAS chart, the patient will choose and record the most appropriate pain rating according to the pain intensity endured.

SECONDARY OUTCOMES:
Radiographic evaluation following the Pulpotomy treatment will be measured | 12 months
  Binary assessment of the radiographs taken after the treatment ( if there is any radiolucent or widening in the lamina sure nor evidence of internal/external pathologic root resorption)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentsitry , Cairo University, Cairo, El Manial, Egypt